CLINICAL TRIAL: NCT03639324
Title: Phase 1 Trial of Rituximab, Idelalisib, and Venetoclax in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (RIVe-CLL/SLL)
Brief Title: Rituximab, Idelalisib, and Venetoclax in Relapsed/Refractory CLL/SLL
Acronym: RIVe-CLL/SLL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15-12310; NCI-2018-01661 (Other: NCI CTRP)
Record Dates: First submitted 2018-08-08; First posted 2018-08-21 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Lymphocytic Leukemia; CLL; Relapsed CLL; Refractory Chronic Lymphocytic Leukemia; Relapsed Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; SLL; Relapsed Small Lymphocytic Lymphoma; Refractory Small Lymphocytic Lymphoma
Keywords: venetoclax; idelalisib; rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: Patients will start on dose level 1 of venetoclax in combination with rituximab and idelalisib, then escalate or de-escalate (if lower dose is available) based upon the estimated probabilities of toxicity from an extension of the continual reassessment method for 2 agents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Combination 1-1 (Experimental): idelalisib + venetoclax
  Interventions: Drug: Dose combination 1-1
- Dose Combination 1-2 (Experimental): idelalisib + venetoclax
  Interventions: Drug: dose combination 1-2
- Dose Combination 1-3 (Experimental): idelalisib + venetoclax
  Interventions: Drug: Dose combination 1-3
- Dose Combination 1-4 (Experimental): idelalisib + venetoclax
  Interventions: Drug: dose combination 1-4
- Sub-Trial Dose Combination 2-1 (Experimental): idelalisib + venetoclax
  Interventions: Drug: Sub-Trial: Dose combination 2-1
- Sub-Trial Dose Combination 2-2 (Experimental): idelalisib + venetoclax
  Interventions: Drug: Sub-Trial: Dose combination 2-2

INTERVENTIONS:
Drug: Dose combination 1-1 — 100 mg QD of idelalisib + 100 mg QD of venetoclax
  Arms: Dose Combination 1-1
Drug: dose combination 1-2 — 100 mg QD of idelalisib + 200 mg QD of venetoclax
  Arms: Dose Combination 1-2
Drug: Dose combination 1-3 — 100 mg BID of idelalisib + 200 mg QD of venetoclax
  Arms: Dose Combination 1-3
Drug: dose combination 1-4 — 150 mg BID of idelalisib + 200 mg QD of venetoclax
  Arms: Dose Combination 1-4
Drug: Sub-Trial: Dose combination 2-1 — 100 mg BID of idelalisib + 100 mg QD of venetoclax
  Arms: Sub-Trial Dose Combination 2-1
Drug: Sub-Trial: Dose combination 2-2 — 150 mg BID of idelalisib + 100 mg QD of venetoclax
  Arms: Sub-Trial Dose Combination 2-2

SUMMARY:
To determine the recommended phase 2 dose (RP2D) of idelalisib and venetoclax in combination with rituximab in patients with relapsed or refractory Chronic lymphocytic leukemia/ Small lymphocytic lymphoma (CLL/SLL) following a lead-in period with idelalisib and rituximab

DETAILED DESCRIPTION:
This phase 1, multicenter, dose-escalation study is designed to find the Recommended Phase 2 Dose (RP2D) of idelalisib and venetoclax in combination with rituximab in patients with relapsed or refractory CLL/SLL and to assess the clinical activity of the combination with rituximab in patients with relapsed or refractory CLL/SLL and to assess the clinical activity of the combination.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years of age. Relapsed or refractory B-cell CLL or biopsy-proven SLL. Treatment required in the opinion of the investigator

Must have had at least one standard treatment with a regimen containing at least one of the following agents/classes of agents; and where specified, must also meet the treatment duration, progression, and/or relapse criteria for that class of agent:

* Fludarabine
* An alkylator (eg, chlorambucil, bendamustine)
* A BTK inhibitor (eg, ibrutinib, acalabrutinib); and must have progressed or relapsed > 6 months after last BTK inhibitor treatment
* An anti-CD20 monoclonal antibody (eg, rituximab, obinutuzumab)
* A BCL-2-family protein inhibitor (eg, venetoclax, navitoclax); and

  * if best response is < CR with BCL-2-family protein inhibitor treatment
  * must have had ≥ 1 year of BCL-2-family protein inhibitor treatment; and
  * must have progressed > 6 months after last BCL-2-family protein inhibitor treatment
  * if best response is CR with BCL-2-family protein inhibitor treatment
  * must have relapsed ≥ 1 year after last BCL-2-family protein inhibitor treatment
* A PI3K inhibitor (eg, idelalisib, duvelisib, TGR-1202, copanlisib, buparlisib); and must have progressed or relapsed > 6 months after last treatment with the PI3K inhibitor (NOTE THAT THIS CRITERION IS NOT APPLICABLE TO 2ND-STEP REGISTRATION)

Prior allogeneic stem cell transplant allowed provided the following criteria are met:

* ≥ 12 months have elapsed since allogeneic transplant
* No current or prior evidence of graft-versus-host disease
* No current requirement for immunosuppressive therapy Prior autologous stem cell transplant allowed provided ≥ 6 months have elapsed since autologous transplant.

Eastern Cooperative Oncology Group performance status of 0, 1, or 2

Adequate bone marrow function as follows:

* Absolute neutrophil count (ANC) ≥ 1,000/mm3 (without support of granulocyte colony stimulating factors)
* Platelets ≥ 50,000/mm3 (untransfused)
* Hemoglobin ≥ 9.0 g/dL

Adequate coagulation, renal, and hepatic function as follows:

* aPTT and PT ≤ 1.2 × upper limit of normal (ULN) for the laboratory
* Calculated creatinine clearance ≥ 50 mL/min as calculated by the standard Cockcroft-Gault equation using age, actual weight, creatinine, and gender
* AST and ALT ≤ 1.5 × ULN for the laboratory
* Bilirubin ≤ 1.5 × ULN for the laboratory. For a woman of childbearing potential (WCBP), a negative serum pregnancy test performed within 7 days prior to initiation of study treatment.

Note: Postmenopausal is defined as any of the following:

* Age ≥ 60 years
* Age < 60 years and amenorrheic for at least 1 year with follicle-stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range
* Bilateral oophorectomy WCBP and male patients must agree to use a medically accepted form of birth control for the duration of study treatment and for at least 1 month following completion of venetoclax and/or idelalisib or 12 months following rituximab, whichever occurs later.

Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

A patient who meets any of the following exclusion criteria is ineligible to participate in the study:

Known histologic transformation from CLL/SLL to an aggressive lymphoma (ie, Richter's transformation).

Known history of drug-induced pneumonitis History of inflammatory bowel disease. Central nervous system involvement Clinically significant infection including active hepatitis B or hepatitis C requiring active treatment, or active CMV infection Known human immunodeficiency virus (HIV) seropositivity. * Note: HIV testing is not required.

Vaccination within 4 weeks prior to initiation of rituximab *Note: Review vaccination status. Patients should, if possible, be brought up-to-date with all immunizations in agreement with current immunization guidelines at least 4 weeks prior to initiating rituximab.•Ongoing requirement for warfarin (due to potential drug-drug interactions that may increase the exposure of warfarin and ensuing complications).

Has received any of the following within 14 days prior to initiation of study treatment:(NOTE THAT THIS CRITERION IS NOT APPLICABLE TO 2ND-STEP REGISTRATION)

* Anti-cancer therapy
* Investigational therapy Has not recovered to ≤ grade 1 toxicity(s) from prior therapy, except for chronic residual toxicities that in the opinion of the investigator are not clinically relevant given the known safety/toxicity profiles of the study regimen (eg, alopecia). (NOTE THAT THIS CRITERION IS NOT APPLICABLE TO 2ND-STEP REGISTRATION) Has not recovered to ≤ grade 1 toxicity(s) from idelalisib and rituximab, except for chronic residual toxicities that in the opinion of the investigator are not clinically relevant given the known safety/toxicity profiles of the study regimen (eg, alopecia). (NOTE THAT THIS CRITERION IS NOT APPLICABLE TO 1ST-STEP REGISTRATION)

Ongoing or planned treatment with any of the following:

* Steroid therapy for anti-neoplastic intent
* Strong or moderate CYP3A inhibitor or inducer, and/or a narrow-therapeutic sensitive substrate
* P-gp inhibitor or narrow-therapeutic sensitive P-gp substrate If any of these agents have been used, patients must be off them for ≥ 1 week before initiation of study treatment.

Prior intolerance to any component of study regimen that, in the opinion of the investigator would preclude study treatment.

A cardiovascular disability status of New York Heart Association Class ≥ II Diagnosis or treatment for another malignancy within 1 year of study registration, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, any in situ malignancy, or low-risk prostate cancer after curative therapy Active liver disease other than lymphoid involvement, inflammatory bowel disease, or Crohn's disease Malabsorption syndrome or other condition that precludes enteral route of administration.

Exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

* Uncontrolled infection (viral, bacterial, or fungal)
* Grade 3 or greater neutropenic fever within 1 week prior to initiation of study treatment Active autoimmune cytopenias (for 2 or more weeks), including autoimmune hemolytic anemia (AIHA) and idiopathic thrombocytopenic purpura.

Pregnancy or breastfeeding Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk, interfere with the patient's participation in the study or hinder evaluation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Find the RP2D of idelalisib and venetoclax in combination with rituximab in patients with relapsed or refractory chronic lymphocytic leukemia/ small lymphocytic lymphoma (CLL/SLL) | 41 Months
  Determine the recommended phase 2 dose of idelalisib and venetoclax in combination with rituximab in patients with relapsed or refractory CLL/SLL following a lead-in period with idelalisib and rituximab.

SECONDARY OUTCOMES:
Safety Evaluation: Determine adverse events (AEs) reported using criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 | 63 Months
  Observed adverse events of treatment with idelalisib and venetoclax in combination with rituximab in patients with relapsed or refractory CLL/ SLL following a lead-in period with idelalisib and rituximab utlizing CTCAE Version 5.0
Determination of cumulative complete response (CR) rate. | 52 Months
  Determine the cumulative CR rate to the study regimen at 7 and 13 months using the 2008 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria.
Summarize the objective response rate. | 52 Months
  Determine the cumulative overall disease response to the study regimen at 7 and 13 months using the 2008 IWCLL criteria.
Minimal residual disease (MRD) rate | 52 Months
  Estimate the rate of undetectable minimal residual disease (MRD) status for idelalisib and venetoclax in combination with rituximab using 4-color flow cytometry in peripheral blood and/or bone marrow for responding patients
Overall Survival Rate | 63 Months
  determine the OS rate (at 24 months following initiation of venetoclax) for idelalisib and venetoclax in combination with rituximab.
Progression Free Survival Rate | 63 Months
  Determine the progression-free survival (PFS) rate (at 24 months following initiation of venetoclax) for idelalisib and venetoclax in combination with rituximab
Pharmacokinetics of the combination of idelalisib and venetoclax. | 7 Years
  Determine the idelalisib and venetoclax plasma concentrations measured at designated time points throughout the study: pre-Tx; C1D1; C1D15; C1D22; C1D29; C3D1; C7D22; C13D222; at DLT (if feasible); at relapse (if feasible)]

CONTACTS AND LOCATIONS:
Overall Officials: Victor Y Yazbek, MD, MS, Principal Investigator — Massey Cancer Center

IPD SHARING:
Plan to Share IPD: No